CLINICAL TRIAL: NCT04203459
Title: Study on the Mechanism of Enhancing the Anti-tumor Effects of Human Chimeric Antigen Receptors T Cells on Pancreatic Cancer by Gut Microbiota Regulation
Brief Title: The Mechanism of Enhancing the Anti-tumor Effects of CAR-T on PC by Gut Microbiota Regulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2019-10-20
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer; Gut Microbiota; CAR-T
Keywords: pancreatic cancer; chimeric antigen receptor T cell; gut microbiota; Acyl-CoA; cholesterol acyltransferase 1; Mesothelin
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — tissue specimens；faeces ；blood；bile .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pancreatic cancer patient: (1) patients with pancreatic cancer confirmed by imaging, pathology and body fluid biopsy, or patients who recovered well one month after operation but still had residual lesions, recurrence or metastasis. ② age ≥ 30 and ≤ 75. ③ no chemotherapy, radiotherapy or targeted drugs were used before admission. ④ patients who had used immunosuppressive drugs, hormones, antibiotics and probiotics one month before admission were excluded. ⑤ patients with HIV positive and active hepatitis B or C infection were excluded. ⑥ exclude the previous history of other malignant tumors or the current combination of other malignant tumors. The patients with serious cardiopulmonary disease and liver and kidney dysfunction were excluded. ⑧ patients with obstructive jaundice were excluded.
- Healthy person: (1) no history of digestive tract diseases, infectious diseases or immune diseases.(2) no history of smoking or drinking.(3) did not take antibiotics and other drugs and probiotics for 1 month before enrollment.

SUMMARY:
Pancreatic cancer (PC) is one of the deadliest diseases of human digestive malignancies. Despite the recent advances in surgery and chemotherapy, the 5-year survival rate of PC continues to be less than 10%. As a promising tumor therapy,Chimeric antigen receptor T cell (CAR-T), however, performed poorly in PC treatment and need to be further updated. In our study, on the basis of our previous research, we use anti-MSLN CAR-T as effector cell and explore the different effects and mechanism of gut microbiota (PC or healthy control) on anti-MSLN CAR-T treatment. Firstly, we detect the differences of gut microbiota and T cell cholesterol metabolism in PC and healthy control by means of 16S-rRNA,PCR, western blot and ELISA; explore the different effects of gut microbiota on the subtype of T cells; and analyze the relationships between intestinal flora composition and T cell cholesterol metabolism or subtype changes by means of Spearman's correlation. Secondly, we also explore the different effects of gut microbiota on the proliferation, migration, subtype, inflammatory cytokines expression and anti-tumor effector function of anti-MSLN CAR-T cells by means of flow cytometry and cytotoxicity assay. Thirdly, we discuss the different expression of cholesterol esterification enzyme 1 (ACAT-1) and other core genes of cholesterol metabolism in anti-MSLN CAR-T. Lastly, we evaluate the effects of different gut microbiota on the treatment of PC by anti-MSLN CAR-T cells in NSG mouse model of subcutaneous PC transplantation and liver metastasis. Through the above experiments, a new theoretical basis is provided in which gut microbiota regulates the subtype and anti-tumor function of anti-MSLN CAR-T by ACAT-1 expression. Furthermore, our findings, which demonstrate the relationship of gut microbiota and CAR-T cell, may be translatable for the treatment of other solid tumors like PC.

ELIGIBILITY:
1. Inclusion criteria and exclusion criteria for the experimental group of this project

Inclusion Criteria:

1. the patients who are confirmed by imaging, pathology and body fluid biopsy to have metastasized pancreatic cancer and can not be cured by operation; or the patients who recover well one month after operation but still have residual focus, recurrence or metastasis.
2. age ≥ 30 and ≤ 75
3. the estimated life span is more than 1 month.
4. Karnofsky score ≥ 60; ECoG ≤ 2
5. the function of important organs: Echocardiography indicated that the ejection fraction of heart was ≥ 50%; ECG showed no obvious abnormality; creatinine clearance rate calculated by Cockcroft Gault formula was ≥ 40ml / min; ALT and AST were ≤ 3 times of normal value; total bilirubin was ≤ 2.0mg/dl; coagulation function: Pt and appt were < 2 times of normal value; arterial oxygen saturation (SpO2) > 92%;Blood routine test: Hgb ≥ 80g / L, ANC ≥ 1 × 109 / L, PLT ≥ 50 × 109 / L.
6. sign the informed consent.

Exclusion Criteria:

1. patients who used immunosuppressive drugs, hormones, antibiotics and probiotics one month before admission.
2. serious active infection.
3. HIV positive, active hepatitis infection.
4. previous history of other malignant tumors. Excluding: Patients with cured skin basal or squamous cell carcinoma and cervical carcinoma in situ at any time before the study; patients with other tumors not listed above but cured by operation only without other further treatment measures and disease-free survival period ≥ 5 years can be included in the study.

(6) patients participating in other clinical trials at the same time. (7) in the opinion of the researcher, the subjects are not suitable to be selected or cannot cooperate to participate in or complete the study.

(8) patients with congenital immunodeficiency. Exclusion criteria

1. patients who had used immunosuppressive drugs, hormones, antibiotics and probiotics in the first month before inclusion.
2. severe active infection.
3. human immunodeficiency virus (HIV) positive, active hepatitis infection.
4. previous history of other malignant tumors. Excluding: patients with cured basal or squamous cell carcinoma of the skin and carcinoma in situ of the cervix at any time prior to the study; Subjects with disease-free survival ≥5 years of other tumors not listed above, which have been cured by surgery only without other further treatment measures, can be included in the study.

(6) patients who also participate in other clinical trials. (7) the investigator considers that the subject is not suitable for inclusion or unable to cooperate in or complete the study.

(8) patients with congenital immune deficiency. (9) a history of myocardial infarction and severe arrhythmia within six months. 2. Inclusion criteria and exclusion criteria for the control group of this project

1. no history of digestive tract diseases, infectious diseases or immune diseases.
2. no history of smoking or drinking.
3. did not take antibiotics and other drugs and probiotics for 1 month before enrollment.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients and Healthy person.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
In vivo experiment: comparison of intestinal microflora and T cell cholesterol metabolism and subtypes between pancreatic cancer patients and healthy people The difference of proportion and the correlation. | from January 2020 to December 2020.
  Fecal and peripheral blood samples were collected from patients with pancreatic cancer and healthy people respectively: (1) through Illumina miseq
  High throughput sequencing technology was used to detect 16S rRNA to analyze the diversity of intestinal flora (α and β diversity), and bioinformatics methods such as random forest and lefse were used to analyze the diversity of flora composition; (2) the difference of cholesterol content in T cells was detected by ELISA; (3) the difference of ACAT-1 expression in T cells was detected by PCR and WB; (4) the difference of ACAT-1 expression in T cells was detected by flow cytometry. The proportion of CD8 +, TNF α +, Th1, Th2, Th17, Treg and other subtypes in T cells was detected by cell analyzer. Furthermore, the correlation between intestinal microflora composition and peripheral blood T cell cholesterol metabolism and subtype difference was determined by Spearman correlation analysis (statistical method).
In vitro experiment: to verify the regulation of intestinal flora on the biological behavior of anti msln car-t in vitro and the role of ACAT-1 in it. | from January 2021 to December 2021.
  In vitro, intestinal flora supernatant of pancreatic cancer and healthy human were co-cultured with anti-msln car-t, respectively, to verify the effect of intestinal flora on biological behavior of anti-msln car-t.To analyze how the metabolism of cholesterol in anti-msln car-t cells, with acat-1 as the key enzyme, participates in the process of regulating the biological behavior of anti-msln car-t by intestinal flora, and preliminarily uncover the relevant mechanism.
Animal model experiment: to verify the ability of intestinal bacteria to control anti msln car-t targeted killing pancreatic cancer cells. | from January 2022 to December 2022.
  Furthermore, the influence of differences in intestinal flora composition between pancreatic cancer and healthy human on anti-msln car-t function was verified in animal models of pancreatic cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No
Personal privacy involved